CLINICAL TRIAL: NCT02757196
Title: Rituximab Plus Short-term Methylprednisolone Versus Standard Dose Methylprednisolone in Newly Diagnosed Participants With Immune Thrombocytopenia (ITP): A Multicenter, Randomized Phase II Study in China
Brief Title: Treatment of ITP With Rituximab and / or Accutane
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Beijing Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ITP Treatment--100
Record Dates: First submitted 2016-04-17; First posted 2016-05-02 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Immune Thrombocytopenia
Keywords: Immune Thrombocytopenia; Rituximab; methylprednisolone
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Rituximab; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rituximab plus methylprednisolone (Experimental): Combination therapy with rituximab （1000mg IV day1, week 3, week 17 , and week 19）plus short-term methylprednisolone (1mg/kg, oral or IV; reduce to 50% of base dose at week 4, then reduce 8mg every 1 week until stopped).
  Interventions: Drug: Rituximab plus methylprednisolone
- Methylprednisolone (Active Comparator): standard dose methylprednisolone alone (1mg/kg, oral or IV; begin to reduce at week 4, reduce 8mg every 2 weeks, then another 8 weeks later reduce 2-4mg every 2-4 weeks).
  Interventions: Drug: methylprednisolone

INTERVENTIONS:
Drug: Rituximab plus methylprednisolone — rituximab （1000mg IV day1, week 3, week 17 , and week 19）
  Other Names: monoclone antibody of cluster of differentiation antigen 20
  Arms: Rituximab plus methylprednisolone
Drug: methylprednisolone — 1mg/kg, oral or IV; begin to reduce at week 4, reduce 8mg every 2 weeks, then another 8 weeks later reduce 2-4mg every 2-4 weeks
  Other Names: intravenous methylprednisolone
  Arms: Methylprednisolone

SUMMARY:
a prospective, multicenter, randomized, open-label, Phase II, two arms interventional trial performed in 5 departments of hematology in China

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, open-label, Phase II, two arms interventional trial performed in 5 departments of hematology in China. The investigators explore the efficacy and safety of Rituximab plus short-term methylprednisolone compare standard dose methylprednisolone in newly diagnosed ITP participants.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically confirmed immune thrombocytopenic purpura (ITP) newly diagnosed
2. Platelet count less than 30×109/L on two occasions or Platelets above 30×109/L combined with bleeding manifestation
3. Subject is ≥ 18 years and ≤80years
4. Subject has signed and dated written informed consent.
5. Fertile patients must use effective contraception during treatment and observational period
6. Negative pregnancy test

Exclusion Criteria:

1. Have an impaired renal function as indicated by a serum creatinine level > 2.0 mg/dL
2. Have an inadequate liver function as indicated by a total bilirubin level > 2.0 mg/dL and/or an aspartate aminotransaminase or alanine aminotransferase level > 3×upper limit of normal
3. Have a New York Heart Classification III or IV heart disease
4. Have a history of severe psychiatric disorder or are unable to comply with study and follow-up procedures
5. Have active hepatitis B or hepatitis C infection
6. Have a HIV infection
7. Have active infection requiring antibiotic therapy within 7 days prior to study entry
8. Are pregnant or lactating women, or plan to become pregnant or impregnated within 12 months of receiving study drug
9. Previous treatment with rituximab
10. Previous splenectomy
11. Had previous or concomitant malignant disease
12. Not willing to participate in the study.
13. Expected survival of < 2 years
14. Intolerant to murine antibodies
15. Immunosuppressive treatment within the last month
16. Connective tissue disease
17. Autoimmune hemolytic anemia
18. Patients currently involved in another clinical trial with evaluation of drug treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Relapse free survival | From date of randomization until the date of relapse or death from any cause, whichever came first, assessed up to 1 year
  Relapse was defined as a drop in platelet count to <30 ×109/L following an initial best response (partial or complete response).

SECONDARY OUTCOMES:
Cumulative response rate | 1 year
  platelet count ≥ 30 x 10^9/L and at least 2-fold increase of the baseline count, confirmed on at least 2 separate occasions at least 7 days apart, and absence of bleeding.
Cumulative complete response rate | 1 year
  platelet count >100 x 10^9/L, confirmed on at least 2 separate occasions at least 7 days apart, and absence of bleeding
Cumulative relapse rate | 1 year
  Time to response (from randomization to the achievement of response)Duration of response (from the initial response to the first relapse)
adverse event/serious adverse event and cumulative rate of bleeding events | 1 year
  adverse event/serious adverse event associated with study drugs and bleeding events

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-jun Huang, Dr, Study Chair — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: No